CLINICAL TRIAL: NCT01693354
Title: Mid-dilution Hemodiafiltration International Randomized Prospective Study on Incident Patients Focused on Outcome
Brief Title: Mid-HDF Randomized Controlled Study on Outcome
Acronym: MILESTONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Antonio Santoro, Professor Antonio Santoro MD, Chief of Nephrology, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MID-INT01
Record Dates: First submitted 2012-09-06; First posted 2012-09-26 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: End Stage Renal Disease
Keywords: dialysis; mortality; cardiovascular stability; inflammation; quality of life
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HF dialysis (Active Comparator): HF (high-flux) dialysis is standard hemodialysis treatment performed by using a high permeability dialyzer instead of a low permeability one.
  Interventions: Device: HF dialysis
- Mid-dilution HDF (Experimental): Mid-dilution is a newly developed hemodiafiltration therapy able to allow a simultaneous pre- and post-dilution infusion.
  Interventions: Device: Mid-dilution HDF

INTERVENTIONS:
Device: Mid-dilution HDF — Mid-dilution HDF is a special, newly developed variant of online HDF which is characterized by a dedicated high-flux hemodialyzer named OLPUR MD able to support simultaneous pre- and post-dilution
  Other Names: OLPUR MD 220; OLPUR MD 190
  Arms: Mid-dilution HDF
Device: HF dialysis — Standard hemodialyzers equipped with high permeability polyphenylene/polyethersulfone membranes
  Other Names: PHYLTHER HF; DIAPES HF
  Arms: HF dialysis

SUMMARY:
The purpose of this study is to determine whether mid-dilution hemodiafiltration is effective in the reduction of the crude mortality risk in patients who have been undergoing renal replacement treatment for less than 1 year. Patients will be randomized since the beginning of the study in two groups: standard HF dialysis and mid-dilution HDF.

DETAILED DESCRIPTION:
It is a matter of fact that in the last decades the Chronic Kidney Disease (CKD) population has widely changed. In Italy, for example, more than 50% of the incident dialysis patients are more than 70 year old, with diabetic and hypertension being the major underlying diseases; moreover a great percentage of the patients starts dialysis with a burden of at least 1-2 comorbidities [1]. Online hemodiafiltration (online HDF) has been recently associated with better patient survival in comparison with standard hemodialysis in two large trials [2,3]; the overall relative risk of mortality was found to be approximately 33% lower in patients treated with online HDF [2,3]. These impressive results were not obtained anyway on the whole population, but in a sub-group analysis. A strong correlation was found between the total convective volume obtained and the mortality risk reduction; HDF was found to be significantly better than standard hemodialysis when a total convective volume of 19-22 L/session (in 4 hours sessions of post-dilution HDF) was achieved.

These results support the importance of the "adequate convective dose" concept in order to improve the patient outcomes especially in frail patients, as recently demonstrated by a large randomised control trial, the MPO study [4], comparing High Flux versus Low Flux dialysis in patients with plasma albumin levels equal to or less than 4 gr/dl ( as a marker of patient comorbidities) and, in a post hoc analysis, in diabetic patients [4].

Mid-dilution HDF is a variant of classical HDF combining simultaneous pre- and post.-dilution in order to maximise middle and large solutes removal.

The MILESTONE study would aim to fully demonstrate for mid-dilution HDF the significant mortality risk reduction observed in the recent mentioned studies.

ELIGIBILITY:
Inclusion Criteria:

* On a thrice/week RRT for at least 3 months
* Dialysis vintage > 3 months
* Signed informed consent
* Blood flow > 300 mL/min

Exclusion Criteria:

* On waiting list for living-donor transplant
* Residual diuresis > 500 mL/day
* Inability, as judget by the investigator, to follow or understand the protocol instructions
* Active neoplastic disease
* Single needle treatment
* Patients with expectancy life lower than 6 months
* Inclusion to other studies
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
crude, all-causes mortality | 5 years
  The primary objective will be assessed by the incidence rate of fatal events

SECONDARY OUTCOMES:
Cardiovascular morbidity | 5 years
  It will be assessed by taking into consideration:
  * Number of hospital admissions related to non fatal major CV events
  * Length of stay during hospitalization
Quality of life and dialysis tolerance evaluated by questionnaire | 1 year
  It will be assessed by taking into consideration:
  - Results of the SF-36 questionnaire given to the patients
Micro-inflammation evaluation | 1 year
  It will be assessed by measuring the pre-dialysis serum levels of:
  IL-6 CR Myoglobin RbP p-cresylsulfate beta2-microglobulin.
  The hospitals' laboratories will be in charge for the sample collection and analysis
Nutrition and anaemia management | 1 year
  It will be assessed by taking in consideration the pre-dialysis serum levels of:
  Hb albumin iron.
  ESAs and iron supplementation will be as well noted in apposite CRF.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Maduell, MD, Study Chair — Hospital Clínic Barcelona, Spain; Vincenzo Panichi, MD, PhD, Study Chair — AUSL 12 Viareggio, Italy; Pedro Aljama, MD, PhD, Study Chair — Hospital Reina Sofia, Cordoba, Spain; Michel Jadoul, MD, PhD, Study Chair — Cliniques Universitaires Saint-Luc, Brussels, Belgium; Philippe Brunet, MD, PhD, Study Chair — Hôpital de la Conception, Marseille, France; Antonio Santoro, MD, Study Chair — AOSP Bologna, Italy
Locations (4):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Hôpital de la Conception, Marseille, France
- Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy
- Hospital Clínic Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Stel VS, van de Luijtgaarden MW, Wanner C, Jager KJ; on behalf of the European Renal Registry Investigators. The 2008 ERA-EDTA Registry Annual Report-a precis. NDT Plus. 2011 Feb;4(1):1-13. doi: 10.1093/ndtplus/sfq191. Epub 2010 Nov 19. PMID 21245934
- [Background] Grooteman MP, van den Dorpel MA, Bots ML, Penne EL, van der Weerd NC, Mazairac AH, den Hoedt CH, van der Tweel I, Levesque R, Nube MJ, ter Wee PM, Blankestijn PJ; CONTRAST Investigators. Effect of online hemodiafiltration on all-cause mortality and cardiovascular outcomes. J Am Soc Nephrol. 2012 Jun;23(6):1087-96. doi: 10.1681/ASN.2011121140. Epub 2012 Apr 26. PMID 22539829
- [Background] Canaud B, Bragg-Gresham JL, Marshall MR, Desmeules S, Gillespie BW, Depner T, Klassen P, Port FK. Mortality risk for patients receiving hemodiafiltration versus hemodialysis: European results from the DOPPS. Kidney Int. 2006 Jun;69(11):2087-93. doi: 10.1038/sj.ki.5000447. PMID 16641921
- [Background] Locatelli F, Martin-Malo A, Hannedouche T, Loureiro A, Papadimitriou M, Wizemann V, Jacobson SH, Czekalski S, Ronco C, Vanholder R; Membrane Permeability Outcome (MPO) Study Group. Effect of membrane permeability on survival of hemodialysis patients. J Am Soc Nephrol. 2009 Mar;20(3):645-54. doi: 10.1681/ASN.2008060590. Epub 2008 Dec 17. PMID 19092122